CLINICAL TRIAL: NCT01412385
Title: A Clinical Study of Immune Globulin Subcutaneous (Human) (IGSC), 20% for the Evaluation of Efficacy, Safety, and Pharmacokinetics in Subjects With Primary Immunodeficiency Diseases
Brief Title: Immune Globulin Subcutaenous (Human), 20%
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170903; 2010-019459-23 (EudraCT Number)
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Patents as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoch 1 (intravenous pre-study treatment) + Epoch 2 (Experimental): Study Epoch 1 (13 weeks): treatment with KIOVIG (once every 3 or 4 weeks, dose as during pre-study period) + Study Epoch 2 (same for all subjects, 51 weeks): treatment with IGSC, 20% (every week, dose to be calculated on the basis of weekly equivalents)
  Interventions: Biological: Immune Globulin Subcutaneous (Human), 20%; Biological: Immune Globulin Intravenous (Human), 10%
- Epoch 1 (subcutaneous pre-study treatment) + Epoch 2 (Experimental): Study Epoch 1 (12 weeks): treatment with SUBCUVIA (once every week or once every two weeks, dose as during pre-study period) + Study Epoch 2 (same for all subjects, 51 weeks): treatment with IGSC, 20% (every week, dose to be calculated on the basis of weekly equivalents)
  Interventions: Biological: Immune Globulin Subcutaneous (Human), 20%; Biological: Human Normal Immunoglobulin (Subcutaneous - Intramuscular Immunoglobulin)

INTERVENTIONS:
Biological: Immune Globulin Subcutaneous (Human), 20% — Subcutaneous infusion (regulated via a pump), Epoch 2 only (all subjects)
  Other Names: IGSC; 20%
Biological: Immune Globulin Intravenous (Human), 10% — Intravenous infusion (regulated via a pump)
  Other Names: GAMMAGARD LIQUID (tradename in the US and Canada); KIOVIG (trademark in Europe)
  Arms: Epoch 1 (intravenous pre-study treatment) + Epoch 2
Biological: Human Normal Immunoglobulin (Subcutaneous - Intramuscular Immunoglobulin) — Subcutaneous infusion (regulated via a pump)
  Other Names: SUBCUVIA
  Arms: Epoch 1 (subcutaneous pre-study treatment) + Epoch 2

SUMMARY:
The purpose of the study is to develop a 20% subcutaneous immunoglobulin treatment option for patients with primary immunodeficiency (PID) diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of a form of primary humoral immunodeficiency involving antibody formation and requiring gammaglobulin replacement, as defined according to the IUIS Scientific Committee 2009, and by diagnostic criteria according to Conley ME, Notarangelo LD, Etzioni A. Diagnostic criteria for primary immunodeficiencies. Clin Immunol 1999; 93:190-197. The diagnosis must be confirmed by the Medical Director prior to enrollment.
* Subject is 2 years or older at the time of screening
* Written informed consent is obtained from either the subject or the subject's legally authorized representative prior to any study-related procedures and study product administration
* Subject has been receiving a consistent dose of IgG over a period of at least 3 months prior to screening at an average minimum dose over that interval equivalent to 300 mg/kg body weight (BW)/4 weeks and a maximum dose equivalent to 1.0 gram/kg BW/4 weeks at a dosing frequency as follows:

  1. intravenously (IV) at mean intervals of approximately 3 or 4 weeks or
  2. subcutaneously (SC) at mean intervals of approximately 1 or 2 weeks
* Subject has a serum trough level of IgG > 5 g/L at screening
* Subject has not had a serious bacterial infection within the 3 months prior to screening
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2
* Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

  1. Persistent alanine aminotransferase (ALT) and aspartate amino transferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
  2. Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] <= 500 /mm3)
* Subject has creatinine clearance (CLcr) value that is < 60% of normal for age and gender
* Subject has been diagnosed with or has a malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix), unless the disease-free period prior to screening exceeds 5 years
* Subject is receiving anti-coagulation therapy or has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) within 12 months prior to screening or a history of thrombophilia
* Subject has abnormal protein loss (protein losing enteropathy, nephrotic syndrome)
* Subject has anemia that would preclude phlebotomy for laboratory studies according to standard practice at the site
* Subject has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IV immunoglobulin, SC immunoglobulin, and/or Immune Serum Globulin (ISG) infusions
* Subject has immunoglobulin A (IgA) deficiency (IgA less than 0.07g/L) and known anti IgA antibodies
* Subject is on preventative (prophylactic) systemic antibacterial antibiotics at doses sufficient to treat or prevent bacterial infections, and cannot stop these antibiotics at the time of screening
* Subject has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening
* Subject has a bleeding disorder or a platelet count less than 20,000/μL, or who, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of subcutaneous therapy
* Subject has total protein >9 g/dL or myeloma, or macroglobulinemia (IgM) or paraproteinemia
* Women of childbearing potential meeting any one of the following criteria

  1. subject presents with a positive pregnancy test
  2. subject is breast feeding
  3. subject intends to begin nursing during the course of the study
  4. subject does not agree to employ adequate birth-control measures (e.g. intrauterine device, diaphragm or condom [for male partner] with spermicidal jelly or foam, or birth control pills/patches) throughout the course of the study
* Subject has participated in another clinical study and has been exposed to an investigational product (IP) or device within 30 days prior to study enrollment (exception: treatment with immunoglobulin pre-study)
* Subject is scheduled to participate in another (non-Baxter) non-observational (interventional) clinical study involving an IP or device during the course of the study
* Subject has severe dermatitis that would preclude adequate sites for safe product administration

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2014-05-13 (Actual); Study Completion 2014-05-13 (Actual)

PRIMARY OUTCOMES:
Acute serious bacterial infection rate defined as the mean number of acute serious bacterial infections per subject per year in the intent-to-treat population | 1 year
  Acute serious bacterial infections will include bacteremia / sepsis, bacterial meningitis, osteomyelitis / septic arthritis, bacterial pneumonia, and visceral abscess, diagnosed according to the Diagnostic Criteria for Serious Acute Bacterial Infections

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Medizinische Universität Wien / AHK Wien (General Hospital Vienna), Universitätsklinik für Kinder- und Jugendheilkunde, Vienna, Austria
- Germany (5):
  - Universitätsklinikum Erlangen, Medizinische Klinik 3, Erlangen
  - University Medical Centre Freiburg, Centre of Chronic Immunodeficiency, Divison of Rheumatology and Clinical Immunology, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Kinderklinik, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Immunologie und Rheumatologie, Hanover
  - Klinikum St. Georg GmbH, Klinik für Kinder- und Jugendmedizin, Leipzig
- Hungary (2):
  - Fővárosi Önkormányzat Egyesített Szent István és Szent László Kórház, Gyermekhematológiai és Őssejt-transzplantációs Osztály, Budapest
  - University of Debrecen, Medical and Health Science Center, Department of Infectious and Pediatric Immunology, Debrecen
- The Queen Silvia Children´s Hospital, Gothenburg, Sweden
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Heart of England NHS Foundation Trust, Immunology Department, Birmingham
  - Addenbrooke´s Hospital, Department of Clinical Immunology, Cambridge
  - Royal London Hospital, Barts and the London NHS Trust, Department of Immunology, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Borte M, Krivan G, Derfalvi B, Marodi L, Harrer T, Jolles S, Bourgeois C, Engl W, Leibl H, McCoy B, Gelmont D, Yel L. Efficacy, safety, tolerability and pharmacokinetics of a novel human immune globulin subcutaneous, 20%: a Phase 2/3 study in Europe in patients with primary immunodeficiencies. Clin Exp Immunol. 2017 Jan;187(1):146-159. doi: 10.1111/cei.12866. Epub 2016 Oct 18. PMID 27613250
- [Derived] Li Z, McCoy B, Engl W, Yel L. Steady-State Serum IgG Trough Levels Are Adequate for Pharmacokinetic Assessment in Patients with Immunodeficiencies Receiving Subcutaneous Immune Globulin. J Clin Immunol. 2021 Aug;41(6):1331-1338. doi: 10.1007/s10875-021-00990-z. Epub 2021 May 26. PMID 34036490
- [Derived] Suez D, Krivan G, Jolles S, Stein M, Gupta S, Paris K, van Hagen PM, Brodszki N, Engl W, Leibl H, McCoy B, Yel L. Safety and tolerability of subcutaneous immunoglobulin 20% in primary immunodeficiency diseases from two continents. Immunotherapy. 2019 Aug;11(12):1057-1065. doi: 10.2217/imt-2019-0057. Epub 2019 Jul 3. PMID 31268374
- [Derived] Paris K, Haddad E, Borte M, Brodszki N, Derfalvi B, Marodi L, Hussain I, Darter A, Engl W, Leibl H, McCoy B, Yel L. Tolerability of subcutaneous immunoglobulin 20%, Ig20Gly, in pediatric patients with primary immunodeficiencies. Immunotherapy. 2019 Apr;11(5):397-406. doi: 10.2217/imt-2018-0088. Epub 2019 Jan 9. PMID 30626238